CLINICAL TRIAL: NCT05602623
Title: Characterizing the Intraocular Scattering at Different Wavelengths
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: CR-6476
Record Dates: First submitted 2022-10-27; First posted 2022-11-02 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Vision, Ocular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (6):
- 770 +/- 9nm/ 830 +/- 15nm/ 900 +/- 15nm (Experimental): Eligible subjects will be randomized to wavelength sequence 770 +/- 9nm/ 830 +/- 15nm/ 900 +/- 15nm. Within each wavelength, subjects will be further randomized to a pupil size sequence (3mm, 4mm, 6mm). Study endpoints will be measured at 3 different pupil sizes.
  Interventions: Device: Adaptive Optics System (AO)
- 770 +/- 9nm/ 900 +/- 15nm/ 830 +/- 15nm (Experimental): Eligible subjects will be randomized to wavelength sequence 770 +/- 9nm/ 900 +/- 15nm/ 830 +/- 15nm. Within each wavelength, subjects will be further randomized to a pupil size sequence (3mm, 4mm, 6mm). Study endpoints will be measured at 3 different pupil sizes.
  Interventions: Device: Adaptive Optics System (AO)
- 830 +/- 15nm/ 770 +/- 9nm/ 900 +/- 15nm (Experimental): Eligible subjects will be randomized to wavelength sequence 830 +/- 15nm/ 770 +/- 9nm/ 900 +/- 15nm. Within each wavelength, subjects will be further randomized to a pupil size sequence (3mm, 4mm, 6mm). Study endpoints will be measured at 3 different pupil sizes.
  Interventions: Device: Adaptive Optics System (AO)
- 830 +/- 15nm/ 900 +/- 15nm/ 770 +/- 9nm (Experimental): Eligible subjects will be randomized to wavelength sequence 830 +/- 15nm/ 900 +/- 15nm/ 770 +/- 9nm. Within each wavelength, subjects will be further randomized to a pupil size sequence (3mm, 4mm, 6mm). Study endpoints will be measured at 3 different pupil sizes.
  Interventions: Device: Adaptive Optics System (AO)
- 900 +/- 15nm/ 830 +/- 15nm/ 770 +/- 9nm (Experimental): Eligible subjects will be randomized to wavelength sequence 900 +/- 15nm/ 830 +/- 15nm/ 770 +/- 9nm. Within each wavelength, subjects will be further randomized to a pupil size sequence (3mm, 4mm, 6mm). Study endpoints will be measured at 3 different pupil sizes.
  Interventions: Device: Adaptive Optics System (AO)
- 900 +/- 15nm/ 770 +/- 9nm/ 830 +/- 15nm (Experimental): Eligible subjects will be randomized to wavelength sequence 900 +/- 15nm/ 770 +/- 9nm/ 830 +/- 15nm. Within each wavelength, subjects will be further randomized to a pupil size sequence (3mm, 4mm, 6mm). Study endpoints will be measured at 3 different pupil sizes.
  Interventions: Device: Adaptive Optics System (AO)

INTERVENTIONS:
Device: Adaptive Optics System (AO) — Subjects will have their higher and lower order aberrations corrected with the AO system.

SUMMARY:
This is a single-site, unmasked, 4-visit, randomized 3x3 cross-over clinical trial to quantify intraocular light scatter in different age groups.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy all the following criteria to be enrolled in the study:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be at least 18 years of age and not greater than 75 years of age at the time of consent.
4. Has had an eye examination within the last two years.
5. The subject's distance vertex corrected spherical equivalent refraction must be in the range of +4.00 D to -6.00 D in each eye.
6. The subject's refractive cylinder must be ≤2.50 D in each eye.
7. The subject must have distance best corrected visual acuity of 20/25 or better in each eye.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

1. Be currently pregnant or lactating.
2. Have any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with their ocular health. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g., hepatitis, tuberculosis).
3. Have any previous, or planned, ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, etc.).
4. Use of any of the following medications within 1 week prior to enrollment: oral retinoid, oral tetracyclines, anticholinergics, oral phenothiazines, oral/inhaled corticosteroids, monoamine oxide inhibitors. See Section 9.1 for further examples.
5. Use of any ocular medication that may interfere with study procedures as determined by the Investigator.
6. Have a history of irregular cornea.
7. Have a history of moderate to severe dry eye.
8. Have Participated in clinical trial within 7 days prior to study enrollment.
9. Be and employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
10. Have any contraindications to pupil dilation.
11. Have any known hypersensitivity, allergic reaction or other contraindication to proparacaine, tropicamide, phenylephrine or sodium fluorescein.
12. Have any allergies to dental mold materials or contraindications to having a dental mold made.
13. Have clinically significant (Grade 3 or greater) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities that may interfere with the study measurements.
14. Have any ocular scars in the central 6 mm of the cornea that may interfere with the study measurement.
15. Have any current ocular infection or inflammation.
16. Intraocular pressure > 21mmHg OD or OS.
17. Ocular angle assessed by Van Herick measurement of grade 2 or less OD or OS.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
Point Spread Function (PSF) for 3mm | up to 2-week follow-up
  Point spread function will be collected in one eye at each Visits 2, 3 and 4 for 3mm pupil size for the assigned wavelength at that visit. The PSF is defined as the way an optical system blurs a point source of light.
Point Spread Function (PSF) for 4 mm | up to 2-week follow-up
  Point spread function will be collected in one eye at each Visits 2, 3 and 4 for 4mm pupil size for the assigned wavelength at that visit. The PSF is defined as the way an optical system blurs a point source of light.
Point Spread Function (PSF) for 6 mm | up to 2-week follow-up
  Point spread function will be collected in one eye at each Visits 2, 3 and 4 for 6mm pupil size for the assigned wavelength at that visit. The PSF is defined as the way an optical system blurs a point source of light.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care Clinical Trial, Study Director — Johnson & Johnson Vision Care
Locations (1):
- University of Houston College of Optometry, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu